CLINICAL TRIAL: NCT01681862
Title: Insights for Community Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Antoinette Schoenthaler, Assistant Professor of Medicine, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HS020982-01A1 (AHRQ); 12-01040 (Other: NYU School of Medicine)
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
Keywords: Hypertension; African American; Personal Health Record; Faith-based Organizations
MeSH Terms: conditions — Hypertension | interventions — Health Records, Personal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personal Health Record (Experimental): Participants data collected during the scheduled blood pressure sessions will be uploaded to the church PHR system. Lay health workers (LHWs) will then have the capability to access the blood pressure readings and health behavior data through the Congregational Dashboard where they can display the information in easy-to-read charts and graphs that highlight the blood pressure trends across the measurements and changes in fruit and vegetable intake, level of physical activity and weight. The registry will also incorporate computerized health education modules through and evidence-based guidelines for blood pressure control and the NHLBI publications "Your Guide to Lowering Blood Pressure" and "Facts about the DASH Eating Plan."
  Interventions: Behavioral: Personal Health Record

INTERVENTIONS:
Behavioral: Personal Health Record — Participants data collected during the scheduled blood pressure sessions will be uploaded to the church PHR system. Lay health workers (LHWs) will then have the capability to access the blood pressure readings and health behavior data through the Congregational Dashboard where they can display the information in easy-to-read charts and graphs that highlight the blood pressure trends across the measurements and changes in fruit and vegetable intake, level of physical activity and weight. The registry will also incorporate computerized health education modules through and evidence-based guidelines for blood pressure control and the NHLBI publications "Your Guide to Lowering Blood Pressure" and "Facts about the DASH Eating Plan."

SUMMARY:
High blood pressure is the number one cause of death for Blacks in the United States. A major reason for the high rates of cardiovascular deaths is poor blood pressure control. Improving blood pressure control leads to large reductions in cardiovascular deaths in Blacks and can be achieved through interventions targeting self-management behaviors. Yet, despite the proven benefits of these interventions, there is little evidence of their role in community-based settings. In NYC, the Department of Health and Mental Hygiene (DOHMH) has developed Keep on Track, a volunteer-run, community program that aims to lower blood pressure of older adults through blood pressure monitoring sessions, brief counseling and health education. With support from DOHMH, lay health workers at faith-based organizations and senior centers take blood pressure readings for community members, record their readings on index cards and provide counseling to support lifestyle change and health care access. However, lay health workers administrating the program report difficulties managing the volume of tracking cards, and express interest in better tools to manage the information. To address this limitation, the primary aim of this study is to test the feasibility of implementing a Personal Health Record (PHR) system in two predominately Black churches in NYC to help lay health workers track changes in blood pressure and health behaviors of the participating congregants. The secondary aims are to evaluate the effect of the PHR system on changes in blood pressure, physical activity, weight loss, fruit and vegetable intake, and number of visits to a primary care physician from baseline to 9 months. The investigators hypothesize that congregants who enroll in the PHR system will have a greater reduction in BP; an increased intake of fruits and vegetables and levels of physical activity; weight loss; and report a great number of visits to their doctor at 9 months.

DETAILED DESCRIPTION:
Poor blood pressure (BP) control is major contributor to the racial disparity in HTN among Blacks; the odds of poor BP control are 40% higher among Blacks as compared to Whites. Improving BP control leads to significant cardiovascular risk reduction in Blacks and can be achieved through evidence-based interventions targeting self-management behaviors that are coordinated with primary care in a "medical neighborhood". Despite the efficacy of these interventions, they are not widely disseminated to community-based settings, or linked as "community resources" to primary care clinics. The challenge for local health departments is to redesign these evidence-based approaches to function at the level of resources and skills available in typical community-based organizations (CBO). Health IT could build the capacity of CBOs to implement evidence-based models, allowing for broader translation of life-saving interventions, and lay a foundation for coordination of care for people with HTN. In New York City, the Department of Health and Mental Hygiene (NYC DOHMH) has developed Keep on Track (KOT) - a volunteer-run program designed to lower BP in older adults through biweekly BP monitoring sessions and health education. With technical and material support from DOHMH, lay health workers (LHW) at senior centers and faith-based organizations take BP readings for community members, record their readings on index cards and provide brief counseling to support lifestyle change and healthcare access. A limitation of the program is the use of paper BP tracking cards, which LHWs find difficult to efficiently review for purposes of targeted outreach and referral. They express interest in alternative tools for information management, which would be more conducive to organized outreach to church members with high BP, to support them in their efforts at lifestyle change and their attempts to gain access to high quality healthcare.

In order to address this important limitation, the investigators will assess the feasibility of implementing a Personal Health Record (PHR) system and Congregational Dashboard customized to support KOT LHWs in two predominately Black churches in NYC to track both individual and aggregate changes in BP and health behaviors among participating congregants. The investigators propose that PHR implementation could improve the capacity of the Health Ministry to manage information and heighten the impact of KOT. Specifically the investigators propose that PHR implementation could improve community-based BP control programs by enabling LHWs to adopt elements of the Chronic Care Model:1) targeted outreach to participating congregants most in need of support for health behavior change; 2) collaborative goal-setting at both the individual and church-level; and 3) empowering members to gain access to healthcare and present physicians with BP tracking reports.

Primary Aim: To assess the feasibility of implementing a customized PHR system to support a church-based BP monitoring program in two predominately Black churches in New York City.

Secondary Aims: To evaluate the effect of implementing the PHR system on:

1. Changes in systolic and diastolic BP from baseline to 9 months
2. Changes in daily servings of fruits and vegetables; level of physical activity; within-participant weight loss; and number of visits to the primary care physician (PCP) from baseline to 9 months

Hypothesis: Congregants who enroll in the PHR system will exhibit a reduction in BP; an increased intake of fruits and vegetables and levels of physical activity; within-participant weight loss; and report a great number of visits to their PCP at 9 months.

Outcomes for the primary and secondary aims will be assessed at the church- and individual-levels. An ongoing formative evaluation will be conducted to identify barriers and facilitators to PHR implementation, and garner suggestions for improvement. Data collected from the formative evaluation will inform necessary system modifications and continuous refinements. A process evaluation will also be conducted with the RE-AIM framework. BP will be assessed with a validated automated BP monitor based on American Heart Association (AHA) guidelines. Health behaviors will be assessed with well-validated self-report measures; weight loss will be estimated as the difference in weight between baseline and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old;
* Are a member of the congregation at one of the participating churches;
* Self-identify as African American/Black and
* Have a diagnosis of HTN (either by self-report or taking at least one antihypertensive medication).

Exclusion Criteria:

* Inability to comply with the study protocol (either self-selected or by indicating during the consent procedures that s/he cannot complete all requested tasks) or
* Has a serious comorbid medical condition (e.g., psychiatric illness, cognitive impairment due to stroke, dementia, Alzheimer's, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | 2 years
  RE-AIM framework and ongoing formative evaluation

SECONDARY OUTCOMES:
Blood pressure | 9 months
  Blood pressure readings will be taken by trained LHWs using a well-validated automated BP monitor. One of the critical factors in this study is the measurement of BP in the church setting. We will select a validated blood pressure monitor that avoids observer bias, can take a series of readings while the patient is seated quietly, and has the capability of uploading the readings into the PHR. In keeping with KOT and AHA guidelines, patients will be seated quietly with an appropriately sized cuff on the non-dominant arm. The device will be programmed to take three readings at one minute intervals, after an initial rest period of five minutes. The average of three readings will be used as the BP measure for each visit.

OTHER OUTCOMES:
Daily servings of fruits and vegetables | 9-months
  Fruit and vegetable intake will be assessed using the 36-item measure developed by Resnicow et al. and validated in a large sample of Black adults participating in the Eat for Life church-based trial. The measure is based on the Health Habits and History Questionnaire and was tailored to foods commonly eaten within the Black population. Participants are asked to indicate number of times that they ate each item in the last seven days and the amount of food (1/2 cup, 1 cup). Portion size is fixed to a medium serving size. The measure will be administered at the baseline and 9-month follow-up visit.
Physical Activity | 9 months
  Physical activity will be assessed with the 7-item International Physical Activity Questionnaire (IPAQ)-short version. The short-IPAQ assesses the amount of health-related vigorous and moderate-intensity physical activity as well as sedentary behaviors in adults over a one week period. The number of hours and minutes per day participants report spending in various types of physical activity is multiplied by the average metabolic equivalent (METs) of each category and summed to calculate energy expenditure as kcal/kg/minutes/week. The IPAQ's reliability and validity is well-established in diverse populations. The measure will be administered at the baseline and 9-month follow-up visit.
Weight loss | 9-months
  Weight will be measured without shoes and with light clothes using a validated digital scale. Measurements will be recorded to the nearest 0.1 kg.
Number of visits to the primary care physician | 9-months
  Number of visits to a PCP will be assessed with a validated single-item developed by the Stanford Research Center. The measure is designed to serve as a proxy for healthcare utilization in the past 6 months and will assist in determining whether the PHR program facilitated coordination of care across the community and clinic settings. Participant that report seeing their PCP will also be asked if they shared their PHR BP tracking reports with the physician. The measure will be administered at the baseline and 9-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, EdD, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - NYC Department of Health and Mental Hygiene, New York, New York
  - NYU School of Medicine, New York, New York